CLINICAL TRIAL: NCT07170397
Title: Effects of a Single Session of Laser Acupuncture Treatment on Blood Pressure and in Hypertension Haemodialysis Patients
Brief Title: Effects of Laser Acupuncture Treatment in Hypertension Haemodialysis Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sinai University (Other)
Responsible Party: Principal Investigator, Amany Gomaa Atiaa, Lecturer in Physical Therapy, Sinai University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SU.REC.2025 (60 H); SU.REC.2025 (60 H) (Other: SinaiU)
Record Dates: First submitted 2025-09-05; First posted 2025-09-12 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Hypertension
Keywords: laser Acupuncture Treatment, Blood Pressure, Hypertension Haemodialysis Patients
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: This expected prospective randomized control trial study will involve 60 haemodialysis patients with hypertension. The patients in the experimental group (E) will subject, medical treatment besides acupuncture laser therapy. Medical treatment will be used in the control group (C). Sleep quality and Blood pressure measurement will be used in the assessment of outcome
Masking Description: This is an open-label study. Both the participants and investigators are aware of the intervention (low-level laser therapy)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Efficacy of of Acupuncture Laser Therapy on Hemodialysis (Active Comparator): Patients receive Acupuncture Laser Therapy
  Interventions: Device: Acupuncture Laser Therapy

INTERVENTIONS:
Device: Acupuncture Laser Therapy — Application of low-level laser therapy to patients with chronic kidney disease to evaluate its effects on pain, circulation, and functional outcomes

SUMMARY:
The purpose of this study is to find the effect of acupuncture laser therapy on Blood Pressure in Hypertension Haemodialysis Patients

DETAILED DESCRIPTION:
In patients with end-stage renal disease (ESRD) receiving dialysis, elevated blood pressure is common and poorly controlled in general. Although volume overload and sodium retention appear to be the main pathogenic mechanism of hypertension in this population, other factors such as increased arterial stiffness, activation of renin-angiotensin-aldosterone system, sleep apnea, activation of sympathetic nervous system, and use of recombinant erythropoietin may be also involved. Acupuncture laser therapy, which uses low-level laser treatment at specific acupuncture points, has shown promise in reducing blood pressure without invasive procedures. However, its specific efficacy in hemodialysis patients remains underexplored, necessitating this research

ELIGIBILITY:
Inclusion Criteria:

* sixty hemodialysis patients undergoing physical therapy treatments will participate in the study. Their mean age will range from (18-65) years old

Exclusion Criteria:

* a failure to take part in more than three light therapy sessions; a kidney transplant; and death

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in systolic and diastolic blood pressure | Baseline and after 4 weeks of low-level laser therapy
  Blood pressure will be measured using a calibrated sphygmomanometer
Blood pressure | Baseline and after 4 weeks of low-level laser therapy
  Blood pressure will be measured using a calibrated sphygmomanometer

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Cairo university- Faculity of physical therapy, Cairo, Cairo Governorate
  - Sinai university- Faculity of physical therapy, El Arish, Sinai

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared

REFERENCES:
- See also: This randomized controlled trial will investigate the effects of low-level laser therapy (LLLT) on blood pressure, functional capacity, and quality of life in patients with chronic kidney disease undergoing hemodialysis. Participants will be randomly ass — https://pubmed.ncbi.nlm.nih.gov/23134313/